CLINICAL TRIAL: NCT00145730
Title: A Multicentre Randomised Placebo-Controlled Trail of Ibuprofen for the Prevention of Ectopic Bone-Related Pain and Disability After Elective Hip Replacement Surgery (HIPAID)
Brief Title: Prevention of Ectopic Bone Related Pain and Disability After Hip Replacement Surgery With Peri-Operative Ibuprofen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Medical Benefits Fund Australia Pty Ltd (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 153712
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2005-09

CONDITIONS: Osteoarthritis, Hip; Arthroplasty, Replacement, Hip; Arthritis, Rheumatoid
Keywords: osteoarthritis hip; arthroplasty; ectopic bone formation; non-steroidal anti-inflammatory drugs; disability
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Ossification, Heterotopic | interventions — Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen

SUMMARY:
The primary aim of this randomised trial is to determine the effects of a short peri-operative course of treatment with a non-steroidal anti-inflammatory drug (NSAID), ibuprofen, on the long-term consequences of ectopic bone formation in patients undergoing elective total hip replacement surgery. The specific hypotheses to be tested at that 6 to 12 months after surgery, patients assigned post-operative ibuprofen will have less self-reported pain and physical disability, greater health-related quality of life and reduced ectopic bone formation compared with those assigned placebo.

DETAILED DESCRIPTION:
Methodology:

The study is a multicentre, randomised, double blind, placebo-controlled trial. 1000 patients undergoing elective total hip replacement surgery from 20 orthopaedic centres in Australia and New Zealand will be assigned to receive either ibuprofen (1200mg daily) or matching placebo in 3 divided doses for 14 days. Study treatment will be started postoperatively on the day of surgery. Patient should not receive any other NSAIDs, apart from low dose aspirin, during the 14-day treatment period, unless such treatment becomes definitely indicated, in which case the study treatment should be withdrawn and open label treatment provided. There will be no other changes to standard care.

Participants:

All patient scheduled for elective total hip replacement surgery, or revision thereof, are potentially eligible unless there is a definite indication for or contraindication to treatment with a NSAID during the 14-day treatment period.

Randomisation:

Randomisation will be performed centrally using a computer-based system that can be accessed 24 hours a day by a toll-free telephone call. A minimisation program will stratify treatment allocation by centre.

Outcomes:

The primary outcome are self-reported pain and physical function, 6 to 12 months after randomisation. Secondary outcomes include health-related quality of life, patients' global assessment, radiographic evidence of ectopic bone.

ELIGIBILITY:
Inclusion Criteria: Patient undergoing elective total hip replacement surgery, or revision thereof -

Exclusion Criteria: A definite indication or contra-indication for treatment with a NSAID during the 14-day study treatment period, in the opinion of the treating clinician.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-02; Study Completion 2004-05

PRIMARY OUTCOMES:
Self-reported pain and physical function (WOMAC)

SECONDARY OUTCOMES:
Health-related quality of life (SF36v2)
Patients' global assessment
Physical performance measures: hip flexion, 50ft walk time, up and go.
Major bleeding events: bleeding from wound > 3 days, evacuation of wound hematoma, hematemesis, melaena, other.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene H Fransen, PhD, MPH, Study Chair — The George Institute, University of Sydney

REFERENCES:
- [Background] Fransen M; HIPAID Management Committee of the HIPAID Collaborative Group. Preventing chronic ectopic bone-related pain and disability after hip replacement surgery with perioperative ibuprofen. A multicenter, randomized, double-blind, placebo-controlled trial (HIPAID). Control Clin Trials. 2004 Apr;25(2):223-33. doi: 10.1016/j.cct.2003.11.008. PMID 15020038
- [Result] Fransen M, Anderson C, Douglas J, MacMahon S, Neal B, Norton R, Woodward M, Cameron ID, Crawford R, Lo SK, Tregonning G, Windolf M; HIPAID Collaborative Group. Safety and efficacy of routine postoperative ibuprofen for pain and disability related to ectopic bone formation after hip replacement surgery (HIPAID): randomised controlled trial. BMJ. 2006 Sep 9;333(7567):519. doi: 10.1136/bmj.38925.471146.4F. Epub 2006 Aug 2. PMID 16885182
- [Derived] Fransen M, Neal B, Cameron ID, Crawford R, Tregonning G, Winstanley J, Norton R; HIPAID Collaborative Group. Determinants of heterotopic ossification after total hip replacement surgery. Hip Int. 2009 Jan-Mar;19(1):41-6. doi: 10.1177/112070000901900108. PMID 19455501